CLINICAL TRIAL: NCT00890929
Title: A Phase 1-2 Study of Azacitidine in Combination With Lenalidomide for Previously Untreated Elderly Patients With Acute Myeloid Leukemia
Brief Title: Phase 1-2 of Azacitidine + Lenalidomide for Previously Untreated Elderly Patients With Acute Myeloid Leukemia (AML)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Principal Investigator, Bruno C. Medeiros, Assistant Professor, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-15611; SU-04242009-2385 (Other: Stanford University); RV-AML-0410 (Other: Celgene Corporation); HEMAML0011 (Other: OnCore)
Record Dates: First submitted 2009-04-28; First posted 2009-04-30 (Estimated); Results first posted 2014-10-20 (Estimated); Last update posted 2018-06-18 (Actual); Status verified 2018-05

CONDITIONS: Acute Myeloid Leukemia (AML); Adult Acute Myeloblastic Leukemia
Keywords: Acute myeloid leukemia; Acute myeloblastic leukemia; AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Lenalidomide; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Azacitidine followed by lenalidomide (Experimental): Dose escalation then dose expansion
  Interventions: Drug: Lenalidomide; Drug: Azacitidine

INTERVENTIONS:
Drug: Lenalidomide — 5 mg, 10 mg, 25 mg, and/or 50 mg of lenalidomide administered PO from day 8 to Day 28 of each cycle
  Other Names: CC-5013; Revlimid
Drug: Azacitidine — 75 mg/m2 Azacitidine administered intravenously (IV) or subcutaneously (SC) for days 1 to 7 of each cycle
  Other Names: 5-azacytidine; Vidaza

SUMMARY:
This study has a phase 1 and a phase 2 component.

In phase 1, the objective is to determine the maximum tolerated dose (MTD) of lenalidomide when after azacitidine.

In phase 2, the objective is to determine the efficacy of the combination treatment.

DETAILED DESCRIPTION:
The treatment regimen in this study is 7 day courses of azacitidine 75 mg/m2 followed by a 21-day courses of lenalidomide. For the primary objective, each 28-day cycle was repeated for a total of up to 6 cycles. Study completion was defined as 18 cycles of treatment, disease progression, or death.

In phase 1, the objective was to determine the maximum tolerated dose (MTD) of lenalidomide 5 mg, 10 mg, 25 mg or 50 mg, when administered after azacitidine.

In phase 2, the objective was to assess the efficacy of MTD lenalidomide administered after azacitidine, in up to six 28-day cycles.

ELIGIBILITY:
Inclusion Criteria

* WHO-confirmed acute myeloid leukemia (AML), except acute promyelocytic leukemia (APL)
* White blood cell count (WBC) at initiation of treatment ≤ 10,000

  ◦If WBC is > 10,000 patients may be started on an appropriate dose of hydroxyurea (to be determined by the investigators), until WBC < 10,000, at which time the hydroxyurea will be discontinued for 24 hours prior to enrollment
* Age ≥ 60 years and not a candidate for allogeneic stem cell transplantation
* Unwilling or unable to receive conventional chemotherapy
* No prior therapy, except supportive care measures such as growth factor support, blood product transfusions, apheresis, or hydroxyurea
* ECOG performance status ≤ 2
* Life expectancy > 2 months
* All study participants must be registered into the mandatory RevAssist® program, and must be willing and able to comply with the requirements of RevAssist
* If a female of childbearing potential (FCBP):

  * Must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10 to 14 days prior to study enrollment and again within 24 hours of prescribing lenalidomide (prescriptions must be filled within 7 days)
  * Must commit to either continued abstinence from heterosexual intercourse or begin two acceptable methods of birth control, one highly effective method and one additional effective method at the same time, at least 28 days before starting lenalidomide.
  * Must also agree to ongoing pregnancy testing.
  * Male partners must use a latex condom during sexual contact, including if the male partners has previously had a successful vasectomy.
* Able to adhere to the study visit schedule and other protocol requirements
* Willing and able to understand and voluntarily sign a written informed consent

Exclusion Criteria

* Relapsed or refractory disease
* Prior therapy with lenalidomide
* History of intolerance to thalidomide or development of erythema nodosum while taking thalidomide or similar drugs
* Known or suspected hypersensitivity to azacitidine or mannitol
* Advanced malignant hepatic tumors
* Concomitant treatment with other anti-neoplastic agents, except hydroxyurea
* Anti-neoplastic treatment less than four weeks prior to enrollment, except hydroxyurea
* Use of any other experimental drug or therapy within 28 days of baseline
* Inability to swallow or absorb drug
* Active opportunistic infection or treatment for opportunistic infection within four weeks of first day of study drug dosing
* New York Heart Association Class III or IV heart failure
* Unstable angina pectoris
* Uncontrolled cardiac arrhythmia
* Uncontrolled psychiatric illness that would limit compliance with requirements
* Known HIV infection
* If female:

  * Pregnant
  * Breast-feeding females, if they do not agree to not breastfeed while taking lenalidomide
* Other medical or psychiatric illness or organ dysfunction or laboratory abnormality which in the opinion of the investigator would compromise the patient's safety or interfere with data interpretation
* Laboratory abnormalities:

  * Creatinine ≥ 1.5 mg/dL
  * Creatinine clearance ≤ 50 mL/min
  * Total bilirubin > 1.5 x institutional upper limit of normal (ULN), except documented Gilbert's syndrome
  * AST > 2.5 x institutional ULN
  * ALT > 2.5 x institutional ULN

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2009-04; Primary Completion 2011-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Carneiro de Medeiros, Principal Investigator — Stanford University; Daniel Aaron Pollyea, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- [Derived] Pollyea DA, Zehnder J, Coutre S, Gotlib JR, Gallegos L, Abdel-Wahab O, Greenberg P, Zhang B, Liedtke M, Berube C, Levine R, Mitchell BS, Medeiros BC. Sequential azacitidine plus lenalidomide combination for elderly patients with untreated acute myeloid leukemia. Haematologica. 2013 Apr;98(4):591-6. doi: 10.3324/haematol.2012.076414. Epub 2012 Dec 14. PMID 23242596
- [Derived] Pollyea DA, Kohrt HE, Gallegos L, Figueroa ME, Abdel-Wahab O, Zhang B, Bhattacharya S, Zehnder J, Liedtke M, Gotlib JR, Coutre S, Berube C, Melnick A, Levine R, Mitchell BS, Medeiros BC. Safety, efficacy and biological predictors of response to sequential azacitidine and lenalidomide for elderly patients with acute myeloid leukemia. Leukemia. 2012 May;26(5):893-901. doi: 10.1038/leu.2011.294. Epub 2011 Oct 28. PMID 22033493

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Azacitidine Followed by Lenalidomide
Started | 45
Consented & Enrolled | 45
Initiated Treatment | 43
Completed | 39
Not Completed | 6
Not completed — Death before treatment | 2
Not completed — Withdrawal by Subject | 3
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Azacitidine Followed by Lenalidomide
Number analyzed (Participants) | 45
Age, Continuous [Median (Full Range); unit: years] | 74 [62 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 28

OUTCOME MEASURES:

1. Primary Outcome: Compete Remission (CR) Rate
Description: Compete Remission (CR) includes subjects with CR but incomplete recovery of blood counts (CRi). CR was assessed according to the European LeukemiaNet (ELN) guidelines, and is defined as the absence of clonal lymphocytes in the peripheral blood.
Time Frame: 12 months
Measure: Number; unit: percentage of subjects
Arm/Group | Azacitidine Followed by Lenalidomide
Number analyzed (Participants) | 43
percentage of subjects | 28

2. Secondary Outcome: 4-week Survival Rate
Description: "Early death" was assessed as death within 28 days of the start of treatment
Time Frame: 28 days
Measure: Number; unit: percentage of subjects remaining alive
Arm/Group | Azacitidine Followed by Lenalidomide
Number analyzed (Participants) | 43
percentage of subjects remaining alive | 83

3. Secondary Outcome: Maximum Tolerated Dose (MTD) of Lenalidomide
Description: The maximum tolerated dose (MTD) of lenalidomide was determined in study phase 1, for use in study Phase 2 (not conducted). The outcome is reported as the dose of lenalidomide that represents the MTD.
Time Frame: 15 months
Population: This outcome only includes results from participants in study Phase 1.
Measure: Number; unit: mg/day lenalidomide (oral)
Arm/Group | Azacitidine Followed by Lenalidomide
Number analyzed (Participants) | 43
mg/day lenalidomide (oral) | 50

4. Secondary Outcome: Remission Duration
Description: Responses and remission were assessed according to the ELN guidelines.
Time Frame: 26 months
Measure: Median (Full Range); unit: weeks
Arm/Group | Azacitidine Followed by Lenalidomide
Number analyzed (Participants) | 43
weeks | 6 [6 to 104]

5. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR includes subjects with CR, CRi, and partial response (PR). Responses were assessed according to the ELN guidelines.
Time Frame: 26 months
Measure: Number; unit: percentage of subjects
Arm/Group | Azacitidine Followed by Lenalidomide
Number analyzed (Participants) | 43
percentage of subjects | 41

6. Secondary Outcome: Overall Survival (OS)
Description: OS from the start of treatment was assessed at a median follow up of 88 weeks from the end of treatment (range, 1-120), and was censored at 1 April 2012.
Time Frame: 88 weeks (median)
Measure: Median (Full Range); unit: weeks
Arm/Group | Azacitidine Followed by Lenalidomide
Number analyzed (Participants) | 43
weeks | 20 [10 to 121]

7. Secondary Outcome: Time to CR
Description: CR includes subjects with CR but incomplete recovery of blood counts (CRi). Responses were assessed according to the ELN guidelines.
Time Frame: 18 weeks
Measure: Median (Full Range); unit: weeks
Arm/Group | Azacitidine Followed by Lenalidomide
Number analyzed (Participants) | 43
weeks | 12 [6 to 18]

8. Secondary Outcome: Time to PR
Description: Responses were assessed according to the ELN guidelines.
Time Frame: 36 weeks
Measure: Median (Full Range); unit: weeks
Arm/Group | Azacitidine Followed by Lenalidomide
Number analyzed (Participants) | 43
weeks | 6 [6 to 36]

9. Secondary Outcome: OS of Responders
Description: OS from the start of treatment of responders (per ELN guidelines) was assessed at a median follow up of 88 weeks from the end of treatment (range, 1-120), and was censored at 1 April 2012.
Time Frame: 88 weeks (median)
Measure: Median (Full Range); unit: weeks
Arm/Group | Azacitidine Followed by Lenalidomide
Number analyzed (Participants) | 43
weeks | 69 [10 to 121]

ADVERSE EVENTS:
Arm/Group | Azacitidine Followed by Lenalidomide
Serious Adverse Events (participants affected / at risk) | 36/43
Other Adverse Events (participants affected / at risk) | 39/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Azacitidine Followed by Lenalidomide (N=43)
Febrile neutropenia (Blood and lymphatic system disorders) | 24 (37)
Blood and lymphatic system disorders - Other, Pancytopenia (Blood and lymphatic system disorders) | 1 (1)
Hemolysis (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Cardiac disorders - Cardiac arrest (Cardiac disorders) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1)
External ear inflammation (Ear and labyrinth disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 1 (1)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Death NOS-AML disease (General disorders) | 2 (2)
Death NOS-Cardiopulmonary arrest (General disorders) | 2 (2)
Death NOS-Chills (General disorders) | 1 (1)
Death NOS-Death (General disorders) | 2 (2)
Death NOS- Thrombocytopenia (General disorders) | 1 (1)
Death NOS-Disease progression (General disorders) | 3 (3)
Death NOS-Hypoxia (General disorders) | 1 (1)
Death NOS-pneumonia (General disorders) | 1 (1)
Death NOS-Sepis (General disorders) | 1 (1)
Death NOS-Terminal Ventricular Tachycardia (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Fever (General disorders) | 2 (2)
Non-cardiac chest pain (General disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Sepsis (Infections and infestations) | 2 (2)
Infections and infestations - Other, Neutropenia (Infections and infestations) | 1 (1)
Platelet count decreased (Investigations) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (2)
Nervous system disorders - Other, high-grade glioblastoma (brain mass) (Nervous system disorders) | 1 (1)
Ischemia cerebrovascular-Acute Stroke (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Respiratory, thoracic and mediastinal disorders - Other, Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypotension (Vascular disorders) | 1 (1)
Vascular disorders - Other, Dieulafoy's lesion (Vascular disorders) | 1 (1)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Azacitidine Followed by Lenalidomide (N=43)
Atrial fibrillation (Cardiac disorders) | 5 (5)
Cardiac disorders - other-Systolic Murmur (Cardiac disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 20 (33)
Diarrhea (Gastrointestinal disorders) | 16 (30)
Dry mouth (Gastrointestinal disorders) | 4 (6)
Dysphagia (Gastrointestinal disorders) | 4 (8)
Hemorrhoids (Gastrointestinal disorders) | 4 (4)
Mucositis oral (Gastrointestinal disorders) | 9 (15)
Nausea (Gastrointestinal disorders) | 23 (50)
Vomiting (Gastrointestinal disorders) | 9 (18)
Edema limbs (General disorders) | 15 (23)
Fatigue (General disorders) | 16 (20)
Fever (General disorders) | 6 (9)
Anorexia (Metabolism and nutrition disorders) | 5 (6)
Injection site reaction (General disorders) | 18 (38)
Urinary tract infection (Infections and infestations) | 5 (6)
Bruising (Injury, poisoning and procedural complications) | 4 (4)
Blood bilirubin increased (Investigations) | 4 (4)
Creatinine increased (Investigations) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (4)
Cognitive disturbance (Nervous system disorders) | 3 (4)
Dizziness (Nervous system disorders) | 5 (6)
Dysgeusia (Nervous system disorders) | 3 (3)
Headache (Nervous system disorders) | 3 (3)
Syncope (Nervous system disorders) | 3 (3)
Tremor (Nervous system disorders) | 5 (6)
Acute kidney injury (Renal and urinary disorders) | 6 (7)
Urinary retention (Renal and urinary disorders) | 4 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 14 (18)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9 (13)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Infections and infestations -- other, Penumonia (Infections and infestations) | 6 (6)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 (6)
Pruritus (Skin and subcutaneous tissue disorders) | 9 (15)
Rash acneiform (Skin and subcutaneous tissue disorders) | 3 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 11 (17)
Neutrophil count decreased (Investigations) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No